CLINICAL TRIAL: NCT02325141
Title: Laparoscopic Sleeve Gasterectomy With or Without Pyloric Sphincter Botulinum Neurotoxin Injection: a Comparative Study
Brief Title: Laparoscopic Sleeve Gasterectomy With or Without Pyloric Botulinum Neurotoxin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Youssef Mohamed, assistant professor of surgery, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MFM201040
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LSG (Active Comparator): patients undergoing laparoscopic sleeve gastrectomy without BTX-A injection into the pyloric sphincter
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- BTX-LSG (Active Comparator): patients undergoing laparoscopic sleeve gastrectomy with BTX-A injection into the pyloric sphincter
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — creation of a gastric tube of 100cc using a stapler.

SUMMARY:
Leakage is the most common complication after laparoscopic sleeve gastrectomy which may amount to 20% in some studies. We hypothesize that Clostridium botulinum neurotoxin A (BTX-A) injection into the pyloric sphincter during the operation may decrease the risk of postoperative gastric leakage.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (LSG) provides similar weight loss and resolution of obesity comorbidities to that of duodenal switch and Roux-en-Y gastric bypass. Inspite of its encouraging results, the pretended feasibility of the operative procedure can be associated with a remarkable operative morbidity. The main reason is gastric leakage from stable line which occurs in about 0-20% of the cases. The main accepted cause of leakage is formation of a high gastric tube pressure. Injection of BTX-A into the pyloric sphincter intraoperative will cause temporal paralysis of pyloric sphincter muscles postoperatively; so the pressure inside the gastric pouch will be decreased abolishing the formation of high pressure tube with subsequent leakage.

ELIGIBILITY:
Inclusion Criteria:

Body mass index >40 or >35 with hypertension or DM

Exclusion Criteria:

Previous bariatric surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
number pf patients developing postoperative gastric leakage | 0ne year

SECONDARY OUTCOMES:
percent of patients with excess weight loss | one year